CLINICAL TRIAL: NCT00892320
Title: A Randomized, Open-label, Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of ER OROS Paliperidone in Healthy Japanese Subjects
Brief Title: A Study of the Effect of Food on the Pharmacokinetics of ER OROS Paliperidone in Healthy Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR004936
Record Dates: First submitted 2008-11-20; First posted 2009-05-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, mood stabilizers, antipsychotics; ER OROS paliperidone
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: ER OROS paliperidone

SUMMARY:
The purposes of this study are to evaluate the effect of food on the pharmacokinetics of extended-release (ER) OROS paliperidone in healthy Japanese adults and to assess the safety and tolerability.

DETAILED DESCRIPTION:
This study was designed as a randomized, open-label, single-center, crossover study to evaluate the effect of food on the pharmacokinetics of extended-release (ER) OROS paliperidone in healthy Japanese adults. Of the 20 Japanese volunteers who are to be enrolled, at least 6 are to be men and 6 are to be women. All volunteers will receive single doses of 3 mg ER OROS paliperidone with and without a standard Japanese breakfast. There will be a 1-week washout between treatments, for a total treatment duration of approximately 2 weeks. Volunteers are to be randomly assigned to 1 of 2 treatment sequence groups (fed and fasted; fasted and fed). The pharmacokinetics of paliperidone will be assessed for 96 hours after each dosing. Safety and tolerability will be monitored throughout the study. Prior to initiating clinical trials in Japan, a food effect study is required to evaluate the effect of food on the pharmacokinetics of ER OROS paliperidone in Japanese adults.

3 mg tablets, single oral dose, once under fasting and once under fed conditions

ELIGIBILITY:
Inclusion Criteria:

* Japanese volunteers must have been born in Japan of Japanese parents and not lived outside of Japan for more than 5 years
* Female volunteers must be surgically sterile, or practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study, have a negative serum beta-HCG pregnancy test at screening and a negative urine pregnancy test on Day -1
* Volunteers must sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
* Volunteers must sign informed consent document for pharmacogenomic testing
* However, participation in the genetic testing component is not mandatory for participation in the remainder of the study
* Volunteers must have a weight as defined by Body Mass Index or Quetelet Index (weight [kg]/height (m)²) within the range of 18.0 - 25.0, extremes included and must be normotensive with supine (5 min) blood pressure between the range of 100-139 mm Hg systolic and 60-89 mm Hg diastolic
* Volunteers must be healthy on the basis of a pre-study physical examination, medical history, electrocardiogram, and the results of blood biochemistry and hematology tests and a urinalysis carried out less than 3 weeks before the first dose. If the results of the biochemistry or hematology tests or the urinalysis testing are not within the laboratory's reference ranges the volunteer can be included only on condition that the investigator judges that the deviations are not clinically significant. For liver function tests (AST, ALT, bilirubin) the values must be within 2 times the upper limit of the normal reference ranges
* Volunteers must smoke less than 10 cigarettes per day and agree not to change smoking habits during the study

Exclusion Criteria:

* Relevant history of any significant and/or unstable cardiovascular, respiratory, neurologic (including seizures or significant cerebrovascular), renal, hepatic, endocrine, psychiatric, or immunologic disorders
* History of any severe preexisting gastrointestinal narrowing (pathologic or iatrogenic)
* Inability to swallow study medication (volunteers may not chew, divide, dissolve, or crush the study medication)
* History or suspicion of alcohol, barbiturate, amphetamine or narcotic abuse
* Drug allergy to risperidone, paliperidone or any of its excipients
* Use of concomitant medication (including vitamins and herbal supplements), except for paracetamol (acetaminophen) and hormonal contraceptives. All other medication must have been stopped at least 14 days before the first dose in the study
* At screening, 2 and 3 minutes after standing, experience a decrease of greater than or equal to 20 mmHg systolic blood pressure, a decrease of greater than or equal to 10 mmHg diastolic blood pressure, or an increase of greater than or equal to 20 beats per minute in heart rate or with symptoms of lightheadedness, dizziness, or fainting upon standing from the supine position
* Positive serology tests for hepatitis B, C or HIV
* Female volunteers that are pregnant, nursing, or planning to become pregnant

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-03; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
to evaluate the effect of food on the pharmacokinetics of extended-release (ER) OROS paliperidone in healthy Japanese adults

SECONDARY OUTCOMES:
to evaluate the safety and tolerability of ER OROS paliperidone in healthy Japanese adults

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the effect of food on the pharmacokinetics of ER OROS paliperidone in healthy Japanese volunteers — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=629&filename=CR004936_CSR.pdf